CLINICAL TRIAL: NCT02521662
Title: A Randomised-controlled Clinical Trial to Evaluate the Effectiveness and Safety of Combining Nicotine Patches With E-cigarettes (With and Without Nicotine) Plus Behavioural Support, on Smoking Abstinence
Brief Title: The Use of Nicotine Patches Together With E-cigarettes (With and Without Nicotine) for Smoking Cessation
Acronym: ASCEND-II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Auckland, New Zealand (Other)
Collaborators: Health New Zealand Ltd, Christchurch, New Zealand (Unknown); Auckland District Health Board (Other Government)
Responsible Party: Principal Investigator, Natalie Walker, Associate Professor of Population Health (Honorary), University of Auckland, New Zealand
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: U1111-1172-9632
Record Dates: First submitted 2015-08-09; First posted 2015-08-13 (Estimated); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Smoking Cessation
Keywords: Electronic Cigarettes; Nicotine Patch; Smoking Cessation
MeSH Terms: conditions — Smoking Cessation; Vaping | interventions — Tobacco Use Cessation Devices; Nicotine Replacement Therapy; Nicotine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Patch (Active Comparator): 21mg nicotine patch daily for 14 weeks (including a 2 week prequit period) plus behavioural support for six weeks post-quit
  Interventions: Drug: Nicotine patch; Behavioral: Behavioural support
- Patch and nicotine-free e-cigarette (Active Comparator): 21mg nicotine patch (daily) and nicotine-free e-cigarette (ad libitum) for 14 weeks (including a 2 week prequit period), plus behavioural support for six weeks post-quit
  Interventions: Drug: Nicotine patch; Device: e-cigarette; Behavioral: Behavioural support
- Patch and nicotine e-cigarette (Active Comparator): 21mg nicotine patch (daily) and nicotine e-cigarette (ad libitum) for 14 weeks (including a 2 week prequit period), plus behavioural support for six weeks post-quit
  Interventions: Drug: Nicotine patch; Device: e-cigarette; Drug: Nicotine; Behavioral: Behavioural support

INTERVENTIONS:
Drug: Nicotine patch — A transdermal patch that slowly releases nicotine into the body through the skin.
  Other Names: Nicotine replacement therapy
Device: e-cigarette — A electronically powered device that delivers to the user an aerosol of propylene glycol and/or glycerine, with or without flavourings and nicotine.
  Other Names: electronic cigarette; electronic nicotine delivery device
  Arms: Patch and nicotine e-cigarette; Patch and nicotine-free e-cigarette
Drug: Nicotine — Nicotine contained in e-liquid (e-juice) used in e-cigarettes
  Other Names: Nicotine liquid
  Arms: Patch and nicotine e-cigarette
Behavioral: Behavioural support — Withdrawal-oriented behavioural support
  Other Names: Smoking cessation behavioural support

SUMMARY:
A randomised trial to determine whether e-cigarettes (with and without nicotine) combined with nicotine patches and behavioural support can assist smokers in remaining abstinent for at least six months.

DETAILED DESCRIPTION:
A pragmatic, double-blind, three-arm randomised controlled trial undertaken in New Zealand to determine whether e-cigarettes combined with nicotine patches can assist smokers in remaining abstinent for at least six months. 1809 smokers who are motivated to quit will be recruited from the community using media advertising and randomly allocated to one of three groups, namely 1) 21mg nicotine patch daily, 2) 21mg nicotine patch daily plus a 'new generation' e-cigarette with no nicotine or 3) 21mg nicotine patch daily plus a 'new generation' e-cigarettes with nicotine. Participants will be instructed to start using the study products two weeks prior to their quit date, and continue for a further 12 weeks after their quit date. Participants will also receive a cessation behavioural support programme consisting of at least six follow-up telephone calls (10-15 minutes each) over the first six weeks. Outcome data will be collected on the participant's set quit date, then one, three, six and (for some but not all) 12 months post-quit date.

ELIGIBILITY:
Inclusion Criteria:

* Smoke and want to quit in the next three months
* Reside in New Zealand
* At least 18 years of age
* Able to provide verbal consent
* Have access to telephone (mobile and/or landline)
* Are prepared to use a nicotine patch or a nicotine patch and e-cigarette together.
* Only one person per household is eligible.

Exclusion Criteria:

* Pregnant women
* Women who are breastfeeding
* Current users of NRT products
* People currently enrolled in another smoking cessation programme or other cessation study
* People who have used an e-cigarette for more than one week in the last year for smoking cessation
* Current users of non-nicotine based cessation therapies (e.g. buproprion, clonidine, nortriptyline or varenicline).
* People who have had a heart attack, stroke or severe angina within the previous two weeks.
* People who self-report a history of severe allergies and/or poorly controlled asthma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1124 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Continuous abstinence (Russell Standard) | Six months post quit date
  Self-report of smoking not more than five cigarettes from the Quit date, supported by biochemical validation (expired air carbon monoxide).

SECONDARY OUTCOMES:
Continuous abstinence | One, three and 12 months post quit date
  Self-report of smoking not more than five cigarettes from the Quit date
7-day point prevalence abstinence | Participant's set quit date, then one, three, six and 12 months post quit date
  Self-report of having smoked no cigarettes (not even a puff) in the past seven days, with biochemical verification at six months only
Number of cigarettes smoked | Participant's set quit date, then one, three, six and 12 months post quit date
  Self-report of number of cigarettes smoked per day (or when smoking for non-daily smokers)
Smoking reduction | Participant's set quit date, then one, three, six and 12 months post quit date
  Defined as reducing consumption by at least 25% (in terms of numbers of cigarettes per day or weight of loose tobacco per day or when smoking for non-daily smokers), at all time points.
Time to relapse | One, three, and six months post quit date
  Time to relapse back to daily smoking from quit date
Withdrawal | Participant's set quit date, then at one month post quit date
  The physical signs and symptoms associated with withdrawal, measured using the Mood and Physical Symptoms Scale (MPSS).
Self-efficacy | Participant's set quit date
  Self-rated chances of quitting, measured on a scale of 1-5 where 1=very low and 5=very high
Use of any other smoking cessation methods/products | Participant's set quit date, then one, three, six and 12 months post quit date
  Participants will be asked whether they used any non-NRT methods of cessation since the last assessment (Yes/No), and if yes, when they started using it, the type they used, and frequency of use.
Serious adverse events | Participant's set quit date, then one, three, six and 12 months post quit date
Cost | Participant's set quit date, then one, three, six and 12 months post quit date
  Cost outcomes will be derived from known costs of the various products include cost per quitter and cost per person reducing their daily cigarette consumption. The tobacco expenditure savings to individual smokers will also be calculated using data on the daily amount smoked prior to quitting and the average price of cigarettes at the time.
Medication compliance | Participant's set quit date, then one and three months post quit date
  How frequently they used their allocated product
Crossover | Participant's set quit date, then one, three, six and 12 months post quit date
  Participants in the patch only arm will be asked whether they accessed and used an e-cigarette (with or without nicotine) during the trial (Yes/No) and at what time during the trial.
Additional e-cigarette support | Participant's set quit date, then one, three, six and 12 months post quit date
  Participants allocated to the e-cigarette groups will be asked whether they accessed any on-line e-cigarette support networks during the trial (Yes/No) and if so what these were (free text), and at what time during the trial.
Dual use | Participant's set quit date, then one, three, six and 12 months post quit date
  Defined as use of both allocated treatment and continued smoking of cigarettes
Continuation of treatment use | Six and 12 months post quit date
  Defined as continued use of allocated treatment after the end of the designated treatment period (12 weeks post-quit).
Perception of their allocated product(s) | Participant's set quit date, then one and three months post quit date
  Participants will be asked what they liked and disliked about their allocated products (free text)
Recommendations | Participant's set quit date, then one and three months post quit date
  Participant's will be asked whether they would recommend their allocated treatment to another smoker who wanted to quit (Yes/No)

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Walker, PhD, Principal Investigator — National Institute for Health Innovation, School of Population Health, University of Auckland
Locations (1):
- National Institute for Health Innovation, University of Auckland, Auckland, North Island, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Walker N, Verbiest M, Kurdziel T, Laking G, Laugesen M, Parag V, Bullen C. Effectiveness and safety of nicotine patches combined with e-cigarettes (with and without nicotine) for smoking cessation: study protocol for a randomised controlled trial. BMJ Open. 2019 Feb 25;9(2):e023659. doi: 10.1136/bmjopen-2018-023659. PMID 30808668
- [Result] Walker N, Parag V, Verbiest M, Laking G, Laugesen M, Bullen C. Nicotine patches used in combination with e-cigarettes (with and without nicotine) for smoking cessation: a pragmatic, randomised trial. Lancet Respir Med. 2020 Jan;8(1):54-64. doi: 10.1016/S2213-2600(19)30269-3. Epub 2019 Sep 9. PMID 31515173
- [Derived] Theodoulou A, Fanshawe TR, Leavens E, Theodoulou E, Wu AD, Heath L, Stewart C, Nollen N, Ahluwalia JS, Butler AR, Hajizadeh A, Thomas J, Lindson N, Hartmann-Boyce J. Differences in the effectiveness of individual-level smoking cessation interventions by socioeconomic status. Cochrane Database Syst Rev. 2025 Jan 27;1(1):CD015120. doi: 10.1002/14651858.CD015120.pub2. PMID 39868569
- [Derived] Hartmann-Boyce J, Theodoulou A, Farley A, Hajek P, Lycett D, Jones LL, Kudlek L, Heath L, Hajizadeh A, Schenkels M, Aveyard P. Interventions for preventing weight gain after smoking cessation. Cochrane Database Syst Rev. 2021 Oct 6;10(10):CD006219. doi: 10.1002/14651858.CD006219.pub4. PMID 34611902